CLINICAL TRIAL: NCT04782596
Title: Transnasal Endoscopic Pituitary Surgery - the Effect of Posterior Nasal Septum Resection on Nasal Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-ENT-Septum
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Pituitary Adenoma
Keywords: pituitary adenoma; nasal functions; posterior nasal septum resection; transnasal approach; endoscopic pituitary surgery
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Intervention Model Description: The study subjects will be randomised into two parallel groups.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-centimeter resection (Experimental): In the study subjects enrolled into this study arm, one-centimetre resection will be used for the transnasal endoscopic pituitary surgery procedure.
  Interventions: Procedure: Posterium nasal septum resection
- Two-centimeter resection (Experimental): In the study subjects enrolled into this study arm, two-centimetre resection will be used for the transnasal endoscopic pituitary surgery procedure.
  Interventions: Procedure: Posterium nasal septum resection

INTERVENTIONS:
Procedure: Posterium nasal septum resection — Posterium nasal septum resection is required to ensure approach during transnasal endoscopic pituitary surgery in patients with pituitary adenoma.

SUMMARY:
The aim of the project is to compare the effect of different extent of resection of the posterior part of the septum on the postoperative nasal functions.

DETAILED DESCRIPTION:
The nasal cavity is used to heat, humidify and purify the air before entering other parts of the respiratory system. Other functions of the nose include in particular olfactory, immune, reflex or sexual functions.

Proper airflow through the nasal cavity is essential for all nasal functions; anatomical or flow changes can significantly affect nasal functions.

Endoscopic transnasal surgical approaches are modern, mini-invasive methods, enabling solution of pathologies in the area of the cranial base, through the nasal cavity. The advantage of this technique is absence of external incisions and scars and significantly better cosmetic effect, these methods also offer very good clarity and illumination of the operating field. Main disadvantage is risk of affecting functions of the nose.

To create a transnasal approach to skull base, it is necessary to perform lateralization of middle turbinates, resection of anterior wall of sphenoidal sinus and resection of posterior part of the nasal septum. These interventions are necessary for a good overview and manipulation in the operated area; however, they can lead to postoperative changes in the physiological functions of the nasal cavity, especially loss of smell, taste, altered airflow through the nasal cavity, mucociliary transport disorders, nasal obstruction, crusting or drying mucous membrane. All these adverse changes significantly affect patient's quality of life.

Larger extent of septal resection allows the surgeon to have a better overview and manoeuvrability in the operated area, which allows sufficient radicality and allows the solution of possible complications. On the other hand, greater resection also means greater interference with the anatomy of the nasal cavity and possible influence on nasal functions.

The aim of the project is to compare the effect of different extent of resection of the posterior part of the septum on the postoperative nasal functions.

Study design:

* all operations will be performed by the same operations team
* prior to surgery, patients will be randomly tossed into two groups according to the extent of resection of the posterior edge of the septum as part of the transsphenoidal approach during cranial base surgery
* group A - Patients will be resected with a posterior 1 cm nasal septum as part of a transsphenoidal approach.
* group B - Patients will be resected with a 2 cm posterior nasal septum as part of a transsphenoidal approach
* if the selected extent of resection is not sufficient during surgery for group A, it will be extended so that the lesion can be safely removed, and patient will be removed from study

Operational procedure:

1. Anemization of the nasal mucosa using strips with diluted adrenaline 1: 1000.
2. Endoscopy of the nasal cavity and identification of important anatomical structures.
3. Lateralization of the middle and upper turbinates, identification of the anterior wall of the sphenoidal sinus and its natural ostium.
4. Apply suction with a marked distance of 1 and 2 cm to the septum and mark the extent of laser resection on the septal mucosa.

   The suction is applied paraseptally to the anterior wall of the sphenoidal sinus at the height of the natural ostium (1.5 cm above the upper edge of the choana), the caudal border of the resection is the height of the upper edge of the choana, the cranial border is the ceiling of the sphenoid.
5. Resection of the septum in the given range.
6. Resection of the anterior wall of the sphenoidal sinus, resection of the intersphenoidal septum.
7. Rest of the operation is identical in both groups of patients (tumour resection, revision of the nasal cavity, nasal tamponade).

   * At preoperative examination and 1 month after surgery, patients will have:
   * endoscopy of the nasal cavity with Lund-Kennedy scoring system (evaluation of oedema, secretion, crust)
   * olfactory examination - test of identification and discrimination with perfumed markers
   * SNOT 22 questionnaire
   * RhinoVAS questionnaire
   * Nose score

Statistical evaluation:

* comparison of nasal functions after cranial base surgery in patients with a range of resection of the posterior edge of the septum 1 cm and 2 cm
* comparison of olfactory before and after surgery in both groups of patients

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* patients with functional pituitary adenoma indicating endoscopic transnasal extirpation of the pituitary adenoma

Exclusion Criteria:

* patients after surgery of the nasal cavity or base of the skull
* patients with nasal disease and PND
* patients with olfactory disorders before surgery
* patients with nasal septal deviation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in nasal endoscopy | 2 months
  Nasal endoscopy will be performed to assess postoperative changes in nasal function (using Lund-Kennedy scoring system)
Changes in sino-nasal outcome test | 2 months
  Sino-nasal outcome test will be used to assess postoperative changes in nasal function (using standardised SNOT 22 questionnaire)
Changes in RhinoVAS questionnaire | 2 months
  RhinoVAS questionnaire will be used to assess postoperative changes in nasal function (using standardised RhinoVAS questionnaire)

SECONDARY OUTCOMES:
Changes in the quality of life | 2 months
  Changes in the quality of life of study subjects will be assessed using standard quality of life measurement tools (e.g. Health-Related Quality of Life - HRQL)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Lubojacký, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. Individual participant data may be provided upon request.

REFERENCES:
- [Background] Alobid I, Ensenat J, Marino-Sanchez F, Rioja E, de Notaris M, Mullol J, Bernal-Sprekelsen M. Expanded endonasal approach using vascularized septal flap reconstruction for skull base tumors has a negative impact on sinonasal symptoms and quality of life. Am J Rhinol Allergy. 2013 Sep-Oct;27(5):426-31. doi: 10.2500/ajra.2013.27.3932. PMID 24119608
- [Background] Rioja E, Bernal-Sprekelsen M, Enriquez K, Ensenat J, Valero R, de Notaris M, Mullol J, Alobid I. Long-term outcomes of endoscopic endonasal approach for skull base surgery: a prospective study. Eur Arch Otorhinolaryngol. 2016 Jul;273(7):1809-17. doi: 10.1007/s00405-015-3853-9. Epub 2015 Dec 19. PMID 26688432
- [Background] Bedrosian JC, McCoul ED, Raithatha R, Akselrod OA, Anand VK, Schwartz TH. A prospective study of postoperative symptoms in sinonasal quality-of-life following endoscopic skull-base surgery: dissociations based on specific symptoms. Int Forum Allergy Rhinol. 2013 Aug;3(8):664-9. doi: 10.1002/alr.21161. Epub 2013 Mar 20. PMID 23520019
- [Background] Bhenswala PN, Schlosser RJ, Nguyen SA, Munawar S, Rowan NR. Sinonasal quality-of-life outcomes after endoscopic endonasal skull base surgery. Int Forum Allergy Rhinol. 2019 Oct;9(10):1105-1118. doi: 10.1002/alr.22398. Epub 2019 Jul 29. PMID 31356005